CLINICAL TRIAL: NCT00171717
Title: Pilot Study of the Conversion From Tacrolimus to Cyclosporine Microemulsion in Liver Transplant Patients Presenting With New Onset Diabetes After the 3rd Month Post-transplant.
Brief Title: Conversion From Tacrolimus to Cyclosporine Microemulsion in Liver Transplant Patients With New Onset Diabetes After the 3rd Month Post-transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLO400AFR04
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Maintenance Liver Transplant Patients With New Onset Diabetes
Keywords: Cyclosporine, liver transplantation, maintenance, diabetes
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: Cyclosporine - cyclosporine microemulsion

SUMMARY:
The trial is conducted in patients who have received a liver transplant, were prescribed tacrolimus to prevent organ rejection and developed diabetes from 3 month post-transplantation onwards. The goal of the trial is to assess the percentage of patients in whom diabetes will resolve 6 month after conversion from tacrolimus to cyclosporine micro-emulsion as measured by a fasting blood glucose < 1,26 g/l without the need of hypoglycemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who have received a first liver transplantation and who are 18 to 70 year old
* Patients who are treated with tacrolimus post-transplant for at least 3 months and for a maximum of 36 months
* Patients without any known diabetes before transplantation and in whom diabetes mellitus was diagnosed for the first time at least 3 months post-transplantation

Exclusion Criteria

* Re-transplantation or multi-organ transplantation,
* Diabetes before the transplantation,
* Type I diabetes mellitus.

Other protocol-defined inclusion / exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-02; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
% of patients whose diabetes resolves 6 months after the conversion (fasting glucose < 1.26 g/L without hypoglycemic treatment).

SECONDARY OUTCOMES:
% of patients whose diabetes has resolved 1 year after the conversion (fasting glucose < 1.26 g/L without hypoglycemic treatment).
% of patients treated with insulin and oral ant diabetics and status of the drug doses 6 months and 1 year after the conversion.
% of patients with HbA1c ≤ 7% 6 months and 1 year after the conversion.
Blood pressure % of patients with a diastolic value ≥ 90 mmHg, mean systolic and diastolic values,
% of patients receiving antihypertensive treatment),
BMI, kidney function (creatinine and creatinine clearance), microalbuminuria, hyperlipidemia, adverse events, serious adverse events, dropouts, at 6 months and at 1 year.
Incidence of acute and chronic rejection treated at 6 months and at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Derived] Lorho R, Hardwigsen J, Dumortier J, Pageaux GP, Durand F, Bizollon T, Blanc AS, Di Giambattista F, Duvoux C. Regression of new-onset diabetes mellitus after conversion from tacrolimus to cyclosporine in liver transplant patients: results of a pilot study. Clin Res Hepatol Gastroenterol. 2011 Jun;35(6-7):482-8. doi: 10.1016/j.clinre.2011.03.008. Epub 2011 May 6. PMID 21530445